CLINICAL TRIAL: NCT03641664
Title: Reducing the Need for Out-of-Home Placements: A Randomized Controlled Trial to Examine the Effects of Family Centered Treatment on Well-Being Outcomes and Public Dollar Costs
Brief Title: FCT Study: Reducing the Need for Out-of-Home Placements
Acronym: 2018-0568
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-0568
Record Dates: First submitted 2018-07-23; First posted 2018-08-22 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Behavior Problem; Mental Disorder; Emotional Problem
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment: Family Centered Treatment (Experimental): Family is offered choice of FCT or Level III out-of-home placement
  Interventions: Behavioral: Family Centered Treatment
- Control: Level III Out of Home Placement (Active Comparator): Family is offered Level III out-of-home placement
  Interventions: Behavioral: Level II or Level III Out of Home Placement

INTERVENTIONS:
Behavioral: Family Centered Treatment — Family Centered Treatment® (FCT) is a promising practice for providing home-based services to families at-risk for their children being removed from home.
  Arms: Treatment: Family Centered Treatment
Behavioral: Level II or Level III Out of Home Placement — Residential care for children with emotional, behavioral, and/or mental health in North Carolina who have experienced a level of dysfunction that makes it impossible to function at an age appropriate level in their own homes or in a lower level of care. These services can be provided in a variety of locations from urban to rural, from facility based to community based and from public sector to private sector. This service provides a structured and supervised environment for the acquisition of skills necessary to enable the child to improve level of functioning to achieve and/or to maintain the most realistic level of independent function where earlier treatment gains are somewhat fragile and the child is subject to regression.
  Arms: Control: Level III Out of Home Placement

SUMMARY:
Does Family Centered Treatment (FCT) result in better youth, family, and cost outcomes, as compared to a Level II or Level III out-of-home placement (OHP)?

The investigators test the hypotheses that among children/youth authorized to a Level II or Level III out-of-home placement, relative to youth who receive such a placement, those who receive FCT will have:

* Better: family functioning and mental/behavioral health outcomes (youth and caregiver).
* Lower probability of: being subject of a child protective services report, entering (or re-entering) foster care, being arrested, being retained in grade, being chronically absent (missing >15 days), dropping out of high school, or receiving an out-of-home placement.
* Lower cost of care.

DETAILED DESCRIPTION:
The goal of this study is to examine the effectiveness of FCT on a number of youth, family, and cost outcomes, as compared to a Level II or Level III out-of-home placement.

Children who are appropriate for Level III service may exhibit the following behaviors:

* Inability to follow directions and conform to structure of school, home or community
* Constant, sometimes violent arguments with caretakers, peers, siblings and/or teachers
* Moderate level of self-injurious behavior, risk taking, sexual promiscuity
* Suicidal actions/history of serious suicidal actions
* Almost daily physical altercations in school, home or community
* Constant verbally aggressive and provocative language
* Frequent and severe property damage
* Probable involvement with the legal system
* Frequent school suspensions
* Moderate to high risk for sexually victimizing others

Typically, children approved for such services are in need of:

* A higher level of supervision and structure than can be provided in a Level II facility;
* Supervision by awake staff during times when the child is sleeping in order to maintain the child;
* A facility that is "staff secure" (i.e., there are no locks, but the child needs a high level of constant supervision to be maintained in the community; and
* Child is only minimally accepting of treatment.

Overall, this service is responsive to the need for intensive, active, therapeutic intervention, which requires a staff secure treatment setting in order to be successfully implemented. This setting has a higher level of consultative and direct service from psychiatrists, psychologists, therapists, medical professionals, etc.

Residential Treatment Level II Service provides a moderate to highly structured and supervised environment. This level of service is responsive to the need for intensive, interactive, therapeutic interventions, which still fall below the level of staff secure/24-hour supervision or secure treatment settings. The staffing structure may include family and program type settings.

A. Program Type The staff is not necessarily awake during sleep time, but must be constantly available to respond to a beneficiary's needs, while beneficiaries are involved in educational, vocational, social or other activities, except for periods of planned respite.

B. Family Type The provider is not necessarily awake during sleep time but must be constantly available to respond to a beneficiary's needs, while beneficiaries are involved in educational, vocational, social or other activities, except for periods of planned respite.

C. Program Type and Family Type Activities

This service in the family or program settings includes the following activities:

1. Individualized and intensive supervision and structure of daily living designed to minimize the occurrence of behaviors related to functional deficits to ensure safety during the presentation of out-of-control behaviors or to maintain an optimum level of functioning.
2. Specific and individualized psychoeducational and therapeutic interventions (e.g., anger management, social skills, family living skills, crisis intervention, etc.)
3. Direct and active intervention in assisting beneficiaries in the process of being involved in and maintaining in naturally occurring community support systems and supporting the development of personal resources (assets, protective factors, etc).

Approximately 750 children/youth will be randomized into one of the two treatments after a Managed Care Organization (MCO) has authorized the OHP request. Birthdays will serve as the method by which children/youth are randomized (e.g., children born on an even numbered day would be randomized into FCT, and children born on an odd numbered day would be randomized into the OHP they were just authorized for). This randomization would occur at the MCO-level, within the Utilization Management division (UM).

Duke-Center for Child & Family Policy (CCFP) staff will approach those families randomized into the OHP (i.e., control group) to participate in the study within a month of the authorization. CCFP and the MCOs will enter into a Business Associate's Agreement (BAA) that will provide CCFP with identified information in order to approach the OHP providers and families about the study.

For those children/youth randomized to receive FCT, MCOs and CCFP staff will work in tandem to notify FCT providers of these potential patients. FCT providers will then approach families about participating in FCT rather than the OHP. They would also recruit the families to participate in the research study, regardless of whether or not the family chooses to participate in FCT. The study would utilize an intent-to-treat design, whereby all families assigned to receive FCT, regardless of whether or not they actually receive the service, will be considered as the "treatment" group in analyses.

ELIGIBILITY:
Inclusion Criteria:

* Participant has been authorized for a level II or level III Out of Home Placement by North Carolina (NC) Division of Medical Assistance
* Youth must have a caregiver and home environment with which to implement FCT,
* Youth must live within a county in NC where FCT service providers implement FCT.

Exclusion Criteria:

* if a youth is currently working with an in-home mental health service provider when the authorization for a Level II or Level III OHP is submitted, that provider cannot be a FCT provider for inclusion into the study
* youth with diagnosed developmental delays or other cognitive impairments will be excluded into the randomization process and recruitment into the longitudinal study.
* Youth for whom the MCO knows that there are current safety concerns which makes them unable to remain in the home with their parent/guardian

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 750 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Family Functioning: General Functioning | baseline, 6 month, 12 months, 18 months
  The Family Assessment Device will be used to measure overall level of family functioning. This subscale ranges from 1 to 4. Higher scores indicate a worse outcome. Both overall functioning and change in functioning will be assessed.
Present Value of FCT compared to Out-of-Home Placement | 1 year
  A cost-benefit analysis will be conducted by calculating the present value in dollars of FCT versus the present value in dollars of out-of-home placement. Behavioral and physical health costs will be measured using claims and encounter data. Higher costs are less desirable than lower costs.
Youth mental health: Child Behavior Checklist(CBCL/YSR), Total Problems | baseline, 6 months, 12 months, 18 months
  The Child Child Behavior Checklist (CBCL)/ Adult Behavior Check List (ABCL)/Youth Self Report (YSR)/Adult Self Report (ASR) are part of The Achenbach System of Empirically Based Assessment (ASEBA) and measures behavioral, emotional, and social behaviors. Respondents rate problem items during the past 6 months as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true".
  The respondent for the CBCL/ABCL is a caregiver. The CBCL is for youth aged 6-18 and the ABCL is for individuals aged 18-59. The respondent for the YSR/ASR are the youth/young adult reporting on him/herself. The CBCL has 113 items, the YSR has 112 items, and the ABCL is 123 items.
  The raw scores are compared with age- and gender-matched controls from a standardization sample; standard scores are derived (mean = 50, standard deviation = 10). Worst score is 80; best score is 30.
  Change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental health: Total Problems | baseline, 6 months, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30.
  Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Present Value of FCT compared to Out-of-Home Placement | 2 years
  A cost-benefit analysis will be conducted by calculating the present value in dollars of FCT versus the present value in dollars of out-of-home placement. Behavioral and physical health costs will be measured using claims and encounter data. Higher costs are less desirable than lower costs.
Present Value of FCT compared to Out-of-Home Placement | 3 years
  A cost-benefit analysis will be conducted by calculating the present value in dollars of FCT versus the present value in dollars of out-of-home placement. Behavioral and physical health costs will be measured using claims and encounter data. Higher costs are less desirable than lower costs.
Present Value of FCT compared to Out-of-Home Placement | 4 years
  A cost-benefit analysis will be conducted by calculating the present value in dollars of FCT versus the present value in dollars of out-of-home placement. Behavioral and physical health costs will be measured using claims and encounter data. Higher costs are less desirable than lower costs.

SECONDARY OUTCOMES:
Family Functioning: Communication | baseline, 6 month, 12 months, 18 months
  The Family Assessment Device will be used to measure how information is exchanged within a family (Communication Subscale). This subscale ranges from 1 to 4. Higher scores indicate a worse outcome. Both overall functioning and change in functioning will be assessed.
Family Functioning: Affective Responsiveness | baseline, 6 month, 12 months, 18 months
  The Family Assessment Device will be used to measure the ability of the family to respond to a range of stimuli with the appropriate quality and quantity of feelings. This subscale ranges from 1 to 4. Higher scores indicate a worse outcome. Both overall functioning and change in functioning will be assessed.
Family Functioning: Problem Solving | baseline, 6 month, 12 months, 18 months
  The Family Assessment Device will be used to measure the family's ability to resolve problems at a level that maintains family functioning. This subscale ranges from 1 to 4. Higher scores indicate a worse outcome. Both overall functioning and change in functioning will be assessed.
Family Functioning: Roles | baseline, 6 month, 12 months, 18 months
  The Family Assessment Device will be used to measure recurrent patterns of behavior by which individuals fulfill family functions. This subscale ranges from 1 to 4. Higher scores indicate a worse outcome. Both overall functioning and change in functioning will be assessed.
Family Functioning: Behavior Control | baseline, 6 month, 12 months, 18 months
  The Family Assessment Device will be used to measure the pattern a family adopts for handling behavior in three types of situations. First, there are physically dangerous situations where the family will have to monitor and control the behavior of its members. Second, there are situations which involve meeting and expressing psychobiological needs or drives such as eating, drinking, sleeping, eliminating, sex and aggression. Finally, there are situations involving interpersonal socializing behavior both among family members and with people outside the family. This subscale ranges from 1 to 4. Higher scores indicate a worse outcome. Both overall functioning and change in functioning will be assessed.
Family Functioning: Affective Involvement | baseline, 6 month, 12 months, 18 months
  The Family Assessment Device will be used to measure the degree to which the family as a whole shows interest in and values the activities and interests of individual family members. This subscale ranges from 1 to 4. Higher scores indicate a worse outcome. Both overall functioning and change in functioning will be assessed.
Youth mental/behavioral health: CBCL/YSR Internalizing Disorder | baseline, 6 month, 12 months, 18 months
  The Child Child Behavior Checklist (CBCL)/ Adult Behavior Check List (ABCL)/Youth Self Report (YSR)/Adult Self Report (ASR) are part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. Respondents rate items (0 = "not true," 1 = "somewhat or sometimes true," 2 = "very true or often true") based on the past 6 months.
  The respondent for the CBCL/ABCL is a caregiver. The CBCL is for youth aged 6-18 and the ABCL is for individuals aged 18-59. The respondent for the YSR/ASR are the youth/young adult reporting on him/herself. The CBCL has 113 items, the YSR has 112 items, and the ABCL is 123 items.
  The raw scores are compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Change in mental health and overall functioning at the various timepoints will be assessed.
Youth mental/behavioral health: CBCL/YSR Externalizing Disorder | baseline, 6 month, 12 months, 18 months
  The Child Child Behavior Checklist (CBCL)/ Adult Behavior Check List (ABCL)/Youth Self Report (YSR)/Adult Self Report (ASR) are part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. Respondents rate items (0 = "not true," 1 = "somewhat or sometimes true," 2 = "very true or often true") based on the past 6 months.
  The respondent for the CBCL/ABCL is a caregiver. The CBCL is for youth aged 6-18 and the ABCL is for individuals aged 18-59. The respondent for the YSR/ASR are the youth/young adult reporting on him/herself. The CBCL has 113 items, the YSR has 112 items, and the ABCL is 123 items.
  The raw scores are compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Change in mental health and overall functioning at the various timepoints will be assessed.
Youth mental/behavioral health: Anxious/Depressed | baseline, 6 month, 12 months, 18 months
  The Child Child Behavior Checklist (CBCL)/ Adult Behavior Check List (ABCL)/Youth Self Report (YSR)/Adult Self Report (ASR) are part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. Respondents rate items (0 = "not true," 1 = "somewhat or sometimes true," 2 = "very true or often true") based on the past 6 months.
  The respondent for the CBCL/ABCL is a caregiver. The CBCL is for youth aged 6-18 and the ABCL is for individuals aged 18-59. The respondent for the YSR/ASR are the youth/young adult reporting on him/herself. The CBCL has 113 items, the YSR has 112 items, and the ABCL is 123 items.
  The raw scores are compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Change in mental health and overall functioning at the various timepoints will be assessed.
Youth mental/behavioral health: Somatic complaints | baseline, 6 month, 12 months, 18 months
  The Child Child Behavior Checklist (CBCL)/ Adult Behavior Check List (ABCL)/Youth Self Report (YSR)/Adult Self Report (ASR) are part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. Respondents rate items (0 = "not true," 1 = "somewhat or sometimes true," 2 = "very true or often true") based on the past 6 months.
  The respondent for the CBCL/ABCL is a caregiver. The CBCL is for youth aged 6-18 and the ABCL is for individuals aged 18-59. The respondent for the YSR/ASR are the youth/young adult reporting on him/herself. The CBCL has 113 items, the YSR has 112 items, and the ABCL is 123 items.
  The raw scores are compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Change in mental health and overall functioning at the various timepoints will be assessed.
Youth mental/behavioral health: Withdrawn Behaviors | baseline, 6 month, 12 months, 18 months
  The Child Child Behavior Checklist (CBCL)/ Adult Behavior Check List (ABCL)/Youth Self Report (YSR)/Adult Self Report (ASR) are part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. Respondents rate items (0 = "not true," 1 = "somewhat or sometimes true," 2 = "very true or often true") based on the past 6 months.
  The respondent for the CBCL/ABCL is a caregiver. The CBCL is for youth aged 6-18 and the ABCL is for individuals aged 18-59. The respondent for the YSR/ASR are the youth/young adult reporting on him/herself. The CBCL has 113 items, the YSR has 112 items, and the ABCL is 123 items.
  The raw scores are compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Change in mental health and overall functioning at the various timepoints will be assessed.
Youth mental/behavioral health: Attention Problems | baseline, 6 month, 12 months, 18 months
  The Child Child Behavior Checklist (CBCL)/ Adult Behavior Check List (ABCL)/Youth Self Report (YSR)/Adult Self Report (ASR) are part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. Respondents rate items (0 = "not true," 1 = "somewhat or sometimes true," 2 = "very true or often true") based on the past 6 months.
  The respondent for the CBCL/ABCL is a caregiver. The CBCL is for youth aged 6-18 and the ABCL is for individuals aged 18-59. The respondent for the YSR/ASR are the youth/young adult reporting on him/herself. The CBCL has 113 items, the YSR has 112 items, and the ABCL is 123 items.
  The raw scores are compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Change in mental health and overall functioning at the various timepoints will be assessed.
Youth mental/behavioral health: Aggressive behavior | baseline, 6 month, 12 months, 18 months
  The Child Child Behavior Checklist (CBCL)/ Adult Behavior Check List (ABCL)/Youth Self Report (YSR)/Adult Self Report (ASR) are part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. Respondents rate items (0 = "not true," 1 = "somewhat or sometimes true," 2 = "very true or often true") based on the past 6 months.
  The respondent for the CBCL/ABCL is a caregiver. The CBCL is for youth aged 6-18 and the ABCL is for individuals aged 18-59. The respondent for the YSR/ASR are the youth/young adult reporting on him/herself. The CBCL has 113 items, the YSR has 112 items, and the ABCL is 123 items.
  The raw scores are compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Change in mental health and overall functioning at the various timepoints will be assessed.
Youth mental/behavioral health: Generalized Anxiety Disorder | baseline, 6 month, 12 months, 18 months
  The Child Child Behavior Checklist (CBCL)/ Adult Behavior Check List (ABCL)/Youth Self Report (YSR)/Adult Self Report (ASR) are part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. Respondents rate items (0 = "not true," 1 = "somewhat or sometimes true," 2 = "very true or often true") based on the past 6 months.
  The respondent for the CBCL/ABCL is a caregiver. The CBCL is for youth aged 6-18 and the ABCL is for individuals aged 18-59. The respondent for the YSR/ASR are the youth/young adult reporting on him/herself. The CBCL has 113 items, the YSR has 112 items, and the ABCL is 123 items.
  The raw scores are compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Change in mental health and overall functioning at the various timepoints will be assessed.
Youth mental/behavioral health: Separation Anxiety Disorder | baseline, 6 month, 12 months, 18 months
  The Child Child Behavior Checklist (CBCL)/ Adult Behavior Check List (ABCL)/Youth Self Report (YSR)/Adult Self Report (ASR) are part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. Respondents rate items (0 = "not true," 1 = "somewhat or sometimes true," 2 = "very true or often true") based on the past 6 months.
  The respondent for the CBCL/ABCL is a caregiver. The CBCL is for youth aged 6-18 and the ABCL is for individuals aged 18-59. The respondent for the YSR/ASR are the youth/young adult reporting on him/herself. The CBCL has 113 items, the YSR has 112 items, and the ABCL is 123 items.
  The raw scores are compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Change in mental health and overall functioning at the various timepoints will be assessed.
Youth mental/behavioral health: Specific Phobia | baseline, 6 month, 12 months, 18 months
  The Child Child Behavior Checklist (CBCL)/ Adult Behavior Check List (ABCL)/Youth Self Report (YSR)/Adult Self Report (ASR) are part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. Respondents rate items (0 = "not true," 1 = "somewhat or sometimes true," 2 = "very true or often true") based on the past 6 months.
  The respondent for the CBCL/ABCL is a caregiver. The CBCL is for youth aged 6-18 and the ABCL is for individuals aged 18-59. The respondent for the YSR/ASR are the youth/young adult reporting on him/herself. The CBCL has 113 items, the YSR has 112 items, and the ABCL is 123 items.
  The raw scores are compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Change in mental health and overall functioning at the various timepoints will be assessed.
Youth mental/behavioral health: Social anxiety disorder | baseline, 6 month, 12 months, 18 months
  The Child Child Behavior Checklist (CBCL)/ Adult Behavior Check List (ABCL)/Youth Self Report (YSR)/Adult Self Report (ASR) are part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. Respondents rate items (0 = "not true," 1 = "somewhat or sometimes true," 2 = "very true or often true") based on the past 6 months.
  The respondent for the CBCL/ABCL is a caregiver. The CBCL is for youth aged 6-18 and the ABCL is for individuals aged 18-59. The respondent for the YSR/ASR are the youth/young adult reporting on him/herself. The CBCL has 113 items, the YSR has 112 items, and the ABCL is 123 items.
  The raw scores are compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Change in mental health and overall functioning at the various timepoints will be assessed.
Youth mental/behavioral health: Somatic symptom disorder | baseline, 6 month, 12 months, 18 months
  The Child Child Behavior Checklist (CBCL)/ Adult Behavior Check List (ABCL)/Youth Self Report (YSR)/Adult Self Report (ASR) are part of The Achenbach System of Empirically Based Assessment (ASEBA)that measures a broad range of behavioral, emotional, and social behaviors. Respondents rate items (0 = "not true," 1 = "somewhat or sometimes true," 2 = "very true or often true") based on the past 6 months.
  The respondent for the CBCL/ABCL is a caregiver. The CBCL is for youth aged 6-18 and the ABCL is for individuals aged 18-59. The respondent for the YSR/ASR are the youth/young adult reporting on him/herself. The CBCL has 113 items, the YSR has 112 items, and the ABCL is 123 items.
  The raw scores are compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Change in mental health and overall functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Adaptive Functioning Scales: Friends | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Adaptive Functioning Scales: Spouse/Partner | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Adaptive Functioning Scales: Family | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Adaptive Functioning Scales: Job | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Adaptive Functioning Scales: Education | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Adaptive Functioning Scales: Personal Strengths | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Syndrome Scales: Anxious/Depressed | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Syndrome Scales: Withdrawn | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Syndrome Scales: Somatic Complaints | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Syndrome Scales: Thought Problems | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Syndrome Scales: Attention Problems | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Syndrome Scales: Aggressive Behavior | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Syndrome Scales: Rule Breaking Behavior | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Syndrome Scales: Intrusive | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Diagnostic and Statistical Manual of Mental Disorders(DSM)-oriented scales-Depressive Symptoms | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: DSM-oriented scales-Anxiety Problems | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: DSM-oriented scales-Somatic Problems | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: DSM-oriented scales-Avoidant Personality Problems | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: DSM-oriented scales-Attention Deficit/Hyperactivity Problems | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: DSM-oriented scales-Antisocial Personality Problems | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Substance Use Scales: Tobacco | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Substance Use Scales: Alcohol | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Substance Use Scales: Drugs | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Substance Use Scales: mean substance use | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Externalizing | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Caregiver mental/Behavioral health: Internalizing | baseline, 6 month, 12 months, 18 months
  The Adult Self Report (ASR) is part of The Achenbach System of Empirically Based Assessment (ASEBA) that measures a broad range of behavioral, emotional, and social behaviors. The ABC is administered in interview format and respondents are asked to rate problem items as 0 for "not true," 1 for "somewhat or sometimes true," and 2 for "very true or often true", based on the past six months.
  The respondent for the ASR is the adult (self). The ASR consists of 126 items.
  The raw scores from the items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are derived with a mean of 50 and a standard deviation of 10. Worst score is 80; best score is 30. Both change in mental health and overall mental health functioning at the various timepoints will be assessed.
Economic Burden: Associated Expenses | Baseline, 6 month, 12 month, 18 month
  The Child and Adolescent Impact Assessment (CAIA) measures the impact that a child or adolescent's symptoms have on the family. The respondent for the CAIA is the parent or caregiver. Respondents will be asked to describe any expenses associated with getting help for their child by responding "there have been no expenses," "there have been expenses, but they have been affordable," or "there have been expenses causing effects on other areas of family budget." A variable will be coded to indicate whether there have been associated expenses (0 = "no expenses," 1 = "expenses but affordable," 2 = "expenses causing effects on other areas of family budget"). Lower expenses are more desirable than higher expenses that are not affordable or effect the family budget.
Economic Burden: Impact on Expenses | Baseline, 6 month, 12 month, 18 month
  The Child and Adolescent Impact Assessment (CAIA) measures the impact that a child or adolescent's symptoms have on the family. The respondent for the CAIA is the parent or caregiver. A series of yes/no questions will ask whether the child's problems have had an impact on family budget for other things, are causing restrictions elsewhere, whether respondent has the savings to cover them, whether respondent has had to work extra hours, and whether the respondent or anyone else has had to take an additional job. A variable will be coded to indicate whether there has been an impact on savings (0 = "absent," 1 = "using savings," 2 = "necessitate cutting back on other expenditures," 3 = "necessitate working additional hours/jobs"). Less impact on family expenses and budget is more desirable than a greater impact.
Economic Burden: Debts | Baseline, 6 month, 12 month, 18 month
  The Child and Adolescent Impact Assessment (CAIA) measures the impact that a child or adolescent's symptoms have on the family. The respondent for the CAIA is the parent or caregiver. Respondents will be asked whether the child's problems have caused them to go into debt to cover expenses or whether they are concerned about being able to pay back expenses. A variable will be coded to indicate whether there are associated debts (0 = "absent," 2 = "incurred debts but envision no serious problems with payback," 3 = "incurred debts and envision will have problems with payback"). Less debt due to expenses is more desirable than incurring debt and having problems paying it back.
Economic Burden: Loss of Income | Baseline, 6 month, 12 month, 18 month
  The Child and Adolescent Impact Assessment (CAIA) measures the impact that a child or adolescent's symptoms have on the family. The respondent for the CAIA is the parent or caregiver. Respondent will be asked whether child's problems have affected family's income. A variable will be coded to indicate whether there has been a loss of income (0 = "absent," 1 = "present"). No loss of income is preferable to any loss of income.
Economic Burden: Impact on Paid Work | Baseline, 6 month, 12 month, 18 month
  The Child and Adolescent Impact Assessment (CAIA) measures the impact that a child or adolescent's symptoms have on the family. The respondent for the CAIA is the parent or caregiver. A series of yes/no questions will be asked to indicate whether child's problems have affected paid work, whether they have lost any time at work, or had to cut down to part-time work, or been unable to work at all, or lost their job. This same series of questions will be asked in relation to both parents and other family members, as applicable. A variable will be coded to indicate whether there has been a loss of income or impact on paid work (0 = "no income lost," 2 = "time lost at work, or hours reduced," 3 = "unable to work or lost job"). No loss of income is preferable to reduced hours or unable to work.
Reported to child protective services | baseline, 6 month, 12 months, 18 months, 2 years, 4 years
  Social service records will be obtained to indicated whether or not a child was referred to child protective services (CPS). This will be scored as yes=1 and no=0 (i.e., range from 0 to 1). Higher values indicate a worse outcome. Both any CPS involvement and repeat use of CPS involvement will be assessed.
Entered Foster care | baseline, 6 month, 12 months, 18 months, 2 years, 4 years
  Social service records will be obtained to indicated whether or not a child entered or re-entered foster care. This will be scored as yes=1 and no=0 (i.e., range from 0 to 1). Higher values indicate a worse outcome. Any entry into foster care care at various time points will be assessed.
Juvenile complaint and/or criminal charges | baseline, 6 month, 12 months, 18 months, 2 years, 4 years
  Whether or not a child was criminally involved will be measured by presence of a juvenile justice complaint and/or adult criminal charge. This information will be obtained through administrative records on juvenile justice, court records and/or corrections records. The range of this will be 0 =no juvenile/criminal record and 1=criminal/juvenile record. Higher scores indicate a worse outcome. A count of the total number of days in which a participant had a juvenile complaint and/or adult charge will also be calculated. Higher scores indicate a worse outcome. Any delinquent or criminal complaints at the various timepoints will be assessed.
Retained in grade | 1 year, 2 years, 3 years, 4 years
  Education records will be used to indicate whether or not an individual repeated a grade in school. This will be scored as 1=retained 0=not retained. Higher values indicate worse outcomes. Any grade retention at the various timepoints will be assessed.
Chronic Absenteeism | 1 year, 2 years, 3 years, 4 years
  Education records will be used to measure whether or not a student was chronically absent from school which will be measured as missed more than 15 days of school (=1) or missed 15 days or fewer days from school. This will be scored as 1=was chronically absent 0=was not chronically absent with higher values indicating a worse outcome. Any chronic absenteeism behavior at the various timepoints will be assessed.
Dropping out of school | 1 year, 2 years, 3 years, 4 years
  Education records will be used to measure whether or not a student dropped out from school (=1). This will be scored as 1=drop out 0=graduated or still in school. Higher values indicate a worse outcome. Whether or not the child has dropped out of school at the various timepoints will be assessed.
Out of home placement | baseline, 6 months, 12 months, 18 months
  The Service Assessment for Children & Adolescents (SACA) will be used to ascertain caregiver reports of whether or not a child had an out of home place for behavioral or emotional or drug or alcohol problems. A series of yes/no questions will ask if their child has stayed overnight in a hospital, treatment center, group or foster home, juvenile justice facility, detention center/prison or jail, or emergency shelter for behavioral, emotional, or drug or alcohol problems. A variable will be created to indicate whether or not the individual was placed out of home (1=yes, 0=0). Higher values indicate worse outcomes. Whether or not the child was placed out of home at the various timepoints will be assessed.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cardinal Innovations Health Care, Charlotte, North Carolina
  - Partners Behavioral Health Management, Elkin, North Carolina